CLINICAL TRIAL: NCT02722746
Title: The Prevention of Hypotension After Epidural Analgesia After Major Surgery by Adding Epinephrine to Infusions to Counteract Sympathectomy: a Double- Blind, Controlled, Randomized, Prospective Dose-finding Study
Brief Title: The Prevention of Hypotension After Epidural Analgesia After Major Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: I. Heermann Anesthesia Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB201600185
Record Dates: First submitted 2016-03-23; First posted 2016-03-30 (Estimated); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Hypotension; Pain
Keywords: Epidural Analgesia
MeSH Terms: conditions — Hypotension; Pain | interventions — Ropivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ropivacaine only Control group (Placebo Comparator): The participants in this group will receive standard anesthesia, epidural analgesia with 0.2% ropivacaine with no epinephrine added during the procedure.
  Interventions: Drug: Ropivacaine
- Ropivacaine + 2 mcg/mL epinephrine (Active Comparator): The participants in this group will receive standard anesthesia (Ropivacaine 0.2%) with the addition of 2mcg/mL of epinephrine during the procedure.
  Interventions: Drug: Ropivacaine; Drug: Epinephrine
- Ropivacaine + 5 mcg/mL epinephrine (Active Comparator): The participants in this group will receive standard anesthesia (Ropivacaine 0.2%) with the addition of 5mcg/mL of epinephrine during the procedure.
  Interventions: Drug: Ropivacaine; Drug: Epinephrine

INTERVENTIONS:
Drug: Ropivacaine — Epidural block infusion with Ropivacaine 0.2% will be provided as the anesthesia per standard of care during the procedure.
  Other Names: Naropin
Drug: Epinephrine — Participants will receive epinephrine in their epidural block infusion during the procedure. The amount of epinephrine provided during the procedure will be based on the group assignment.
  Other Names: Adrenalin
  Arms: Ropivacaine + 2 mcg/mL epinephrine; Ropivacaine + 5 mcg/mL epinephrine

SUMMARY:
Epidural analgesia via continuous epidurally infused local anesthetic agent (LA) is widely and very successfully used routinely for perioperative pain control in patients undergoing major orthopedic and abdominal surgery since 1928. The choice currently depends on the preference of the APS physician in charge of the case. A frequent unwanted side effect of epidural block is hypotension due to the epidurally injected LA blocking the sympathetic nerves and thus the patient's response to hypotension, which is usually due to hypovolemia and/or an unopposed parasympathetic (via the vagus nerve) nervous system. The purpose of this research study is to see if adding epinephrine, to the epidural anesthetic will decrease possible side effects, such as low blood pressure, and lead to a better effect of the epidural anesthetic.

DETAILED DESCRIPTION:
Participants undergoing epidural analgesia to treat perioperative pain associated with major surgery will be approached for their willingness to participate in the study. Participants undergoing major thoracic, abdominal, or orthopaedic surgery for whom thoracic or lumbar epidural block would be indicated and planned for intraoperative and postoperative analgesia as per the University of Florida Acute Pain Service (APS) usual and routine practice will be included in this study.

All participants will receive a standardized continuous epidural block at the appropriate level for the planned surgery by the APS physicians in the block room that day. For the standardized continuous epidural block, placement will be confirmed with loss of resistance technique (LORA), wave form analysis or nerve stimulation.

Participants will be randomly allocated by computer-generated randomization to one of four groups. This will be a quintuple blinded prospective study. The anesthesiologist managing the intraoperative anesthesia, the anesthesiologists (APS) placing the blocks and following the participants on the floors, the research nurse taking the measurement, the surgeons, nor the participants will be aware of what combination of drugs are used for the epidural block infusion.

The three groups will consist of:

1. Group A (Ropivacaine 0.2% infusion; Control group)
2. Group B (Ropivacaine 0.2% + 2 mcg/mL epinephrine)
3. Group C (Ropivacaine 0.2% + 5 mcg/mL epinephrine)

ELIGIBILITY:
Inclusion Criteria:

* undergoing epidural analgesia to treat perioperative pain associated with major surgery
* undergoing major thoracic surgery
* undergoing major abdominal surgery
* undergoing major orthopaedic surgery

Exclusion Criteria:

* sepsis
* acute trauma
* coagulopathy
* preoperative hemodynamic instability
* symptomatic coronary artery disease
* patients from the ICU whose tracheas were intubated for any cause
* allergies to medications in the protocol
* primary or secondary block failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2017-10-04 (Actual); Study Completion 2018-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olga C. Nin, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nin OC, Boezaart A, Giordano C, Hughes SJ, Parvataneni HK, Reina MA, Schirmer A, Vasilopoulos T. Pilot epinephrine dose-finding study to counter epidural-related blood pressure reduction. Reg Anesth Pain Med. 2025 Nov 5;50(11):901-906. doi: 10.1136/rapm-2024-105406. PMID 38991714

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ropivacaine Only Control Group | Ropivacaine + 2 mcg/mL Epinephrine | Ropivacaine + 5 mcg/mL Epinephrine
Started | 23 | 21 | 22
Completed | 15 | 16 | 16
Not Completed | 8 | 5 | 6
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Protocol Violation | 8 | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropivacaine Only Control Group | Ropivacaine + 2 mcg/mL Epinephrine | Ropivacaine + 5 mcg/mL Epinephrine | Total
Number analyzed (Participants) | 15 | 16 | 16 | 47
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.5 (14.2) | 52.8 (16.8) | 57.3 (14.5) | 58.7 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 7 | 22
  Male | 7 | 9 | 9 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Type of Surgery [Count of Participants; unit: Participants]
  Abdominal | 9 | 7 | 12 | 28
  Orthopedia | 6 | 9 | 4 | 19
Type of Block [Count of Participants; unit: Participants]
  Lumbar | 6 | 9 | 4 | 19
  Thoracic | 9 | 7 | 12 | 28

OUTCOME MEASURES:

1. Primary Outcome: Changes Between the 3 Groups Assessed by Blood Pressure Measurement
Description: Hypotension will be assessed by systolic blood pressure (SBP) > 20% below the baseline preoperative measurements and acquired before the epidural or any sedation has been administered and the intra-operative period. The median time to end of intraoperative period was 2:37 (hours:min), ranging from 0:53 to 7:30.
Time Frame: Change from baseline to end of the intra-operative period
Measure: Count of Participants; unit: Participants
Arm/Group | Ropivacaine Only Control Group | Ropivacaine + 2 mcg/mL Epinephrine | Ropivacaine + 5 mcg/mL Epinephrine
Number analyzed (Participants) | 15 | 16 | 16
Participants
  Hypotension | 5 | 2 | 3
  No Hypotension | 10 | 14 | 13
Statistical Analysis 1: Comparison: Ropivacaine Only Control Group vs Ropivacaine + 2 mcg/mL Epinephrine; Test type: Superiority; p = 0.165, Z-test for proportions; percent difference = 20.8, 95% CI 2-sided [-8.9 to 47.3]
Statistical Analysis 2: Comparison: Ropivacaine Only Control Group vs Ropivacaine + 5 mcg/mL Epinephrine; Test type: Superiority; p = 0.353, Z-test for proportions; percent difference = 14.4, 95% CI 2-sided [-15.9 to 42.2]

2. Secondary Outcome: Changes Between the 3 Groups Assessed by the Spread of Local Anesthetic (Block) Effect
Description: Spread of local anesthetic (block) effect as tested by sensitivity to cold recorded every hour postoperatively and every 8 hours for the subsequent 72 hours after discharge from the PACU. Cold was applied to dermatomes (i.e. segments/areas of skin primarily assoicated with one spinal nerve), then sensitivty to cold was recorded to determine spread of block across spinal segments.
Time Frame: Preop, post anesthesia care unit (PACU), Post-op Da 1 (POD 1, 72 hours after discharge from PACU)
Measure: Median (Inter-Quartile Range); unit: dermatomes
Arm/Group | Ropivacaine Only Control Group | Ropivacaine + 2 mcg/mL Epinephrine | Ropivacaine + 5 mcg/mL Epinephrine
Number analyzed (Participants) | 14 | 12 | 14
dermatomes
  PACU | 8 [6 to 9] | 11 [8 to 13] | 9 [7 to 10]
  Pre-op | 10 [9 to 12] | 9 [7 to 11] | 7 [5 to 10]
  POD 1 | 7 [7 to 10] | 6 [6 to 10] | 8 [6 to 12]
Statistical Analysis 1: Comparison: Ropivacaine Only Control Group vs Ropivacaine + 2 mcg/mL Epinephrine vs Ropivacaine + 5 mcg/mL Epinephrine; For PACU spread; Test type: Superiority; p = 0.06, Kruskal-Wallis
Statistical Analysis 2: Comparison: Ropivacaine Only Control Group vs Ropivacaine + 2 mcg/mL Epinephrine vs Ropivacaine + 5 mcg/mL Epinephrine; For Pre-op spread; Test type: Superiority; p = 0.22, Kruskal-Wallis
Statistical Analysis 3: Comparison: Ropivacaine Only Control Group vs Ropivacaine + 2 mcg/mL Epinephrine vs Ropivacaine + 5 mcg/mL Epinephrine; For POD 1; Test type: Superiority; p = 0.74, Kruskal-Wallis

3. Secondary Outcome: Changes Between the 3 Groups Assessed by Ambulation After Surgery
Description: Ambulation on post-op day 1, post-op day 2 and post-op day 3, will be recorded by distance ambulated per 24-hour period, calculating mean ambulation in feet per day
Time Frame: From post-operative (post-op) day 1 to post-op day 3
Measure: Mean (95% Confidence Interval); unit: feet per day
Arm/Group | Ropivacaine Only Control Group | Ropivacaine + 2 mcg/mL Epinephrine | Ropivacaine + 5 mcg/mL Epinephrine
Number analyzed (Participants) | 13 | 14 | 13
feet per day | 125.5 [58.3 to 192.7] | 90.2 [25.5 to 155.0] | 139.1 [71.9 to 206.3]
Statistical Analysis 1: Comparison: Ropivacaine Only Control Group vs Ropivacaine + 2 mcg/mL Epinephrine vs Ropivacaine + 5 mcg/mL Epinephrine; Test type: Superiority; p = 0.551, ANOVA

4. Secondary Outcome: Changes Between the 3 Groups Assessed by Opioid Usage
Description: Opioid usage data will be recorded and converted to morphine equivalents and averaged for day 0, and post-op days 1, 2, and 3 per group.
Time Frame: From day of surgery (0) to post-op day 3
Population: Putcome was only recorded for patients that remained hospitalized and does not included those that were discharged, thus lower numbers in later POD measurement.
Measure: Mean (95% Confidence Interval); unit: Morphine milligram equivalents
Arm/Group | Ropivacaine Only Control Group | Ropivacaine + 2 mcg/mL Epinephrine | Ropivacaine + 5 mcg/mL Epinephrine
Number analyzed (Participants) | 15 | 16 | 16
Morphine milligram equivalents
  POD 0 | 27.2 [1.7 to 52.7] | 40.4 [16.7 to 64.2] | 14.9 [-7.4 to 37.2]
  POD 1 | 41.9 [16.2 to 67.6] | 65.1 [39.4 to 90.8] | 28.3 [4.2 to 53.1]
  POD 2: number analyzed (Participants) | 10 | 12 | 13
  POD 2 | 28.0 [4.9 to 51.1] | 47.5 [26.4 to 68.6] | 26.7 [6.4 to 47.0]
  POD 3: number analyzed (Participants) | 8 | 4 | 6
  POD 3 | 45.5 [6.8 to 84.6] | 19.8 [-35 to 74.6] | 26.9 [-17.8 to 71.7]
Statistical Analysis 1: Comparison: Ropivacaine Only Control Group vs Ropivacaine + 2 mcg/mL Epinephrine vs Ropivacaine + 5 mcg/mL Epinephrine; Test type: Superiority; p = 0.349, Mixed Models Analysis

5. Secondary Outcome: Changes Between the 3 Groups Assessed by Opioid-related Side Effects
Description: Side effects such as pruritus, nausea/vomiting, and respiratory depression (defined as respiratory rate less than 10 breaths per minute of oxygen saturation more than 7 points lower that the patients preoperative value on room air) will be recorded.
Time Frame: From day of surgery (0) to post-op day 3
Population: Outcome was was recorded up until POD 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Ropivacaine Only Control Group | Ropivacaine + 2 mcg/mL Epinephrine | Ropivacaine + 5 mcg/mL Epinephrine
Number analyzed (Participants) | 15 | 16 | 16
Participants
  Pruritis | 1 | 5 | 1
  Nausea/vomiting | 5 | 8 | 9
  Respiratory Depression | 12 | 12 | 14
Statistical Analysis 1: Comparison: Ropivacaine Only Control Group vs Ropivacaine + 2 mcg/mL Epinephrine vs Ropivacaine + 5 mcg/mL Epinephrine; For Pruritis; Test type: Superiority; p = 0.18, Fisher Exact
Statistical Analysis 2: Comparison: Ropivacaine Only Control Group vs Ropivacaine + 2 mcg/mL Epinephrine vs Ropivacaine + 5 mcg/mL Epinephrine; For Nausea/Vomiting; Test type: Superiority; p = 0.44, Fisher Exact
Statistical Analysis 3: Comparison: Ropivacaine Only Control Group vs Ropivacaine + 2 mcg/mL Epinephrine vs Ropivacaine + 5 mcg/mL Epinephrine; For Respirartory Depression; Test type: Superiority; p = 0.74, Fisher Exact

6. Secondary Outcome: Changes Between the 3 Groups Assessed by Fluid Balance
Description: 24 hour intake and output for, the first 72 hours (up until POD 3) to assess fluid balance, reported as median intake and output per day (in milliliters per day).
Time Frame: From post-op day 1 to post-op day 3
Population: change was measured earlier if discharge if before 72 hours.
Measure: Median (Full Range); unit: milliliters per day
Arm/Group | Ropivacaine Only Control Group | Ropivacaine + 2 mcg/mL Epinephrine | Ropivacaine + 5 mcg/mL Epinephrine
Number analyzed (Participants) | 15 | 16 | 16
milliliters per day
  Drain Output | 164 [0 to 1635] | 305 [109 to 458] | 315 [0 to 2162]
  IV Intake | 2428 [872 to 4185] | 1300 [700 to 3615] | 1843 [512 to 3859]
  PO Intake | 542 [0 to 2147] | 308 [0 to 1483] | 477 [13 to 743]
  Urine Output | 1921 [550 to 2483] | 1600 [276 to 2300] | 1100 [100 to 2250]

7. Secondary Outcome: Changes Between the 3 Groups Assessed by Length of Hospitalization
Description: Length of hospitalization, recorded as median days
Time Frame: post-op period, up until discharge
Measure: Median (Full Range); unit: days
Arm/Group | Ropivacaine Only Control Group | Ropivacaine + 2 mcg/mL Epinephrine | Ropivacaine + 5 mcg/mL Epinephrine
Number analyzed (Participants) | 15 | 16 | 16
days | 4 [1 to 11] | 2 [1 to 12] | 2 [1 to 17]

8. Secondary Outcome: Changes Between the 3 Groups Assessed by Days to Return to Oral Intake Status
Description: Return to oral intake (PO) status, recorded in median days
Time Frame: post-op period, up until discharge
Measure: Median (Full Range); unit: days
Arm/Group | Ropivacaine Only Control Group | Ropivacaine + 2 mcg/mL Epinephrine | Ropivacaine + 5 mcg/mL Epinephrine
Number analyzed (Participants) | 15 | 16 | 16
days | 1 [0 to 4] | 1 [0 to 5] | 1 [0 to 4]

9. Secondary Outcome: Changes Between the 3 Groups Continously Measured Cardiovascular Outcomes - Blood Pressure
Description: Changes in systolic blood pressure (SBP) , diastolic blood pressure (DBP), mean arterial blood pressure (MAP) assesed by area-under-the-curve calculated using pre-op as reference value. Measures were summarized across four time intervals, preoperative, intraoperative, PACU, and transfer to floor, with these intervals as x-axis for AUC
Time Frame: Change across preoperative, intraoperative, Post Anesthesia Care Unit (PACU), and transfer to floor (up to 72 hours)
Measure: Mean (95% Confidence Interval); unit: mmHg * hours
Arm/Group | Ropivacaine Only Control Group | Ropivacaine + 2 mcg/mL Epinephrine | Ropivacaine + 5 mcg/mL Epinephrine
Number analyzed (Participants) | 15 | 16 | 16
mmHg * hours
  SBP | -9.6 [-33.7 to 14.5] | -5.0 [-8.6 to 18.7] | -4.5 [-23.2 to 1421]
  DBP | -0.3 [-13.9 to 13.2] | -6.1 [-17.1 to 5.0] | -8.2 [-18.8 to 2.4]
  MAP | 6.4 [-9.3 to 22.2] | -6.4 [-21.0 to 8.1] | -11.6 [-26.7 to 3.4]
Statistical Analysis 1: Comparison: Ropivacaine Only Control Group vs Ropivacaine + 2 mcg/mL Epinephrine vs Ropivacaine + 5 mcg/mL Epinephrine; For SBP; Test type: Superiority; p = 0.524, ANOVA
Statistical Analysis 2: Comparison: Ropivacaine Only Control Group vs Ropivacaine + 2 mcg/mL Epinephrine vs Ropivacaine + 5 mcg/mL Epinephrine; For DBP; Test type: Superiority; p = 0.585, ANOVA
Statistical Analysis 3: Comparison: Ropivacaine Only Control Group vs Ropivacaine + 2 mcg/mL Epinephrine vs Ropivacaine + 5 mcg/mL Epinephrine; For MAP; Test type: Superiority; p = 0.199, ANOVA

10. Secondary Outcome: Differences Between the 3 Groups Assessed by Pain
Description: Pain measured by and visual analog pain score on the Defense and Veterans Pain Rating Scale. This scale ranges from 0 to 10, with higher scores indicating greater pain. Pain scores were average within in 12-hour time interval for comparison.
Time Frame: Measured at 12-hour intervals for first 48 hours postopoerative
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ropivacaine Only Control Group | Ropivacaine + 2 mcg/mL Epinephrine | Ropivacaine + 5 mcg/mL Epinephrine
Number analyzed (Participants) | 15 | 16 | 16
units on a scale
  0-12 hours | 3.5 [2.4 to 4.7] | 2.5 [1.4 to 3.7] | 4.3 [3.2 to 5.5]
  12-24 hours | 4.4 [2.9 to 5.8] | 3.9 [2.5 to 5.3] | 3.9 [2.3 to 5.5]
  24-36 hours | 4.3 [2.9 to 5.8] | 4.3 [3.0 to 5.6] | 3.5 [2.3 to 4.7]
  36-48 hours | 3.0 [1.5 to 4.6] | 3.7 [2.2 to 5.1] | 3.6 [2.4 to 4.9]
Statistical Analysis 1: Comparison: Ropivacaine Only Control Group vs Ropivacaine + 2 mcg/mL Epinephrine vs Ropivacaine + 5 mcg/mL Epinephrine; Test type: Superiority; p = 0.231, Mixed Models Analysis

11. Secondary Outcome: Changes Between the 3 Groups Continously Measured Cardiovascular Outcomes - Respiratory Rate
Description: Changes in respiratory rate (RR) assesed by area-under-the-curve (AUC) calculated using pre-op as reference value. Measures were summarized across four time intervals, preoperative, intraoperative, PACU, and transfer to floor, with these intervals as x-axis for AUC
Time Frame: Change from preoperative, intraoperative, Post Anesthesia Care Unit (PACU), and transfer to floor (up to 72 hours)
Measure: Mean (95% Confidence Interval); unit: breaths/min * hours
Arm/Group | Ropivacaine Only Control Group | Ropivacaine + 2 mcg/mL Epinephrine | Ropivacaine + 5 mcg/mL Epinephrine
Number analyzed (Participants) | 15 | 16 | 16
breaths/min * hours | -10.2 [-13.7 to 6.7] | -4.2 [-8.3 to .02] | -3.6 [-6.7 to -0.4]
Statistical Analysis 1: Comparison: Ropivacaine Only Control Group vs Ropivacaine + 2 mcg/mL Epinephrine vs Ropivacaine + 5 mcg/mL Epinephrine; Test type: Superiority; p = 0.016, ANOVA

12. Secondary Outcome: Changes Between the 3 Groups Continously Measured Cardiovascular Outcomes - Heart Rate
Description: Changes in heart rate (HR) assesed by area-under-the-curve calculated using pre-op as reference value. Measures were summarized across four time intervals, preoperative, intraoperative, PACU, and transfer to floor, with these intervals as x-axis for AUC
Time Frame: Change across preoperative, intraoperative, Post Anesthesia Care Unit (PACU), and transfer to floor (up to 72 hours)
Measure: Mean (95% Confidence Interval); unit: beats/min * hours
Arm/Group | Ropivacaine Only Control Group | Ropivacaine + 2 mcg/mL Epinephrine | Ropivacaine + 5 mcg/mL Epinephrine
Number analyzed (Participants) | 15 | 16 | 16
beats/min * hours | 17.3 [-33.5 to 22.2] | -2.1 [-11.3 to 7.2] | 0.9 [-9.6 to 11.4]
Statistical Analysis 1: Comparison: Ropivacaine Only Control Group vs Ropivacaine + 2 mcg/mL Epinephrine vs Ropivacaine + 5 mcg/mL Epinephrine; Test type: Superiority; p = 0.055, ANOVA

13. Secondary Outcome: Changes Between the 3 Groups Continously Measured Cardiovascular Outcomes - Oxygen Saturation
Description: Changes in oxygen saturation (SpO2), and heart rate (HR) assesed by area-under-the-curve calculated using pre-op as reference value. Measures were summarized across four time intervals, preoperative, intraoperative, PACU, and transfer to floor, with these intervals as x-axis for AUC
Time Frame: Change across preoperative, intraoperative, Post Anesthesia Care Unit (PACU), and transfer to floor (up to 72 hours)
Measure: Mean (95% Confidence Interval); unit: % saturation * hours
Arm/Group | Ropivacaine Only Control Group | Ropivacaine + 2 mcg/mL Epinephrine | Ropivacaine + 5 mcg/mL Epinephrine
Number analyzed (Participants) | 15 | 16 | 16
% saturation * hours | 11.5 [-17.9 to 40.9] | 1.8 [-4.6 to 8.2] | 0.3 [-2.5 to 3.2]
Statistical Analysis 1: Comparison: Ropivacaine Only Control Group vs Ropivacaine + 2 mcg/mL Epinephrine vs Ropivacaine + 5 mcg/mL Epinephrine; Test type: Superiority; p = 0.567, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse events were recording across postoperative period until dishcarge
Arm/Group | Ropivacaine Only Control Group | Ropivacaine + 2 mcg/mL Epinephrine | Ropivacaine + 5 mcg/mL Epinephrine
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 12/15 | 14/16 | 14/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ropivacaine Only Control Group (N=15) | Ropivacaine + 2 mcg/mL Epinephrine (N=16) | Ropivacaine + 5 mcg/mL Epinephrine (N=16)
Pruritis (Skin and subcutaneous tissue disorders) | 2 | 5 | 1
Nausea/Vomiting (Gastrointestinal disorders) | 5 | 8 | 9
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 12 | 12 | 14 — RR less than 10bmp or Sa)2 sat >7pts below baseline

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-09): https://cdn.clinicaltrials.gov/large-docs/46/NCT02722746/Prot_SAP_000.pdf